CLINICAL TRIAL: NCT02921490
Title: Molecular and Magnetic Resonance Imaging Biomarkers of Facet Joint Pain of the Lumbar Spine With PET/MRI
Brief Title: FDG PET/MRI Evaluation of Facet Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vance Lehman, M.D. , Assistant Professor of Radiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-001228
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/MR recipients (Experimental): All recruited patients will undergo FDG PET/MR of the lumbar spine as the single arm of the study.
  Interventions: Device: FDG PET/MR examination.

INTERVENTIONS:
Device: FDG PET/MR examination. — All recruited patients will undergo an FDG PET examination focused on the lumbar spine.

SUMMARY:
Chronic pain incurs over half a trillion dollars in lost productivity (healthcare, lost wages, etc) annually. The most common source is low back pain (LBP), often from facet joints. The clinical evaluation of facet joints is challenging and anatomic imaging findings of facet joint; degenerative change; correlate poorly with pain. Therefore, it is difficult to select appropriate candidate patients/facet joints to treat. Misguided percutaneous treatment can cost thousands of dollars per session and delay diagnoses. Very limited retrospective information suggests that high grade peri-facet MRI signal change correlates to the side of LBP. However, this has not fully characterized the imaging findings and has not correlated to expert clinical exam/percutaneous response, precluding robust and meaningful clinical impact. Minimal retrospective data concludes inflammatory changes can be identified on FDG-PET exams, but the evidence of correlation to patient pain is lacking. Limited DWI exists for inflammatory spondyloarthropathies and myopathies, but is also lacking.

This is an exploratory study investigating the utility of FDG PET activity and MRI signal change around facet joints in the clinical management of low back pain. This study will help determine if such imaging biomarkers could change clinical management. Additionally, this will provide data that will be vital to planning a larger prospective study evaluating the ability of imaging biomarkers to predict response to comparison medial branch blocks and RF ablation for treatment of facet joint pain.

DETAILED DESCRIPTION:
10 patients with a clinical suspicion of at least 60% likelihood that low back pain arises from the lumbar facet joints will be recruited in clinic. The clinicians will rate the likelihood clinically of facet joint origin of pain and will assign a theoretical treatment plan based on initial clinical impression. They will indicate which facet joints, if any, they would refer for percutaneous treatment. The patients will undergo and FDG PET/MRI of the lumbar spine with IV gadolinium. The MRI signal change and enhancement of the lumbar facet joints will be graded by 2 radiologists blinded to the clinical data. The FDG PET scan activity of the facet joints will be graded by two nuclear medicine radiologists blinded to the clinical information. The clinicians will then be segmentally unblended to the imaging data as follows: 1. facet joints with high grade MRI signal change, 2. facet joints with any MRI signal change, 3. facet joints with high grade PET activity, and 4. facet joints with any PET activity. At each of these 4 steps, the clinician will indicate if this information would have the potential to alter clinical care (assuming that the imaging biomarker in question would be a surrogate for inflammation and pain) and if the information is concordant to the clinical impression. The clinical course of each patients will be followed for 1 year after undergoing the PET/MRI examination.

ELIGIBILITY:
Eligibility criteria - inclusion:

1. Male and female patients over the age of 50-100 years with clinically suspected facetogenic low back pain.
2. Patients must be considered to have at least a 60% chance of having facet joints as the major source of low back pain based on overall clinical impression.
3. All patients will undergo a standardized clinical exam by an experienced physical medicine and rehabilitation clinician to confirm clinical suspicion of axial low back pain.
4. Patients with either unilateral or bilateral axial low back pain may be enrolled.

Eligibility criteria - exclusion:

1. Pregnancy
2. Prior lumbar back surgery
3. History of endovascular repair of abdominal aortic aneurysm or other postoperative change likely to introduce imaging artifact to the lumbar spine
4. Suspected spine infection
5. Known osseous metastatic or other osseous malignancy
6. Facet joint percutaneous treatment within the past 2 months
7. History of major lumbar spine trauma
8. Inability to provide own consent
9. Claustrophobia, cardiac pacemaker/wires in place, any absolute contraindication to MRI
10. Impaired renal function indicated by a GFR less than 30
11. Gadolinium allergy
12. Highly radiosensitive medical conditions
13. Patients who are unable to lay quietly for 60 minutes of imaging

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vance T Lehman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PET/MR Recipients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 63 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Number of patients with back pain [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Facet Joint High Grade FDG Activity Concordance to Pain
Description: Concordance of high grade FDG scores with clinical impression
Time Frame: 2 years
Measure: Number; unit: concordance correlation coefficient
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
concordance correlation coefficient | 0.10

2. Primary Outcome: Facet Joint All Grades of FDG Activity Concordance to Pain
Description: Number/percentage of subjects (reported in sides, with two sides (Left or Right) per patient) for whom any grade (any evidence of increased FDG activity) of FDG scores are in concordance with clinical impression
Time Frame: 2 years
Population: The measure is best reported in sides, which is 2 sides per patient. 10 patients with 20 sides.
Measure: Number; unit: sides (left or right)
Units Other Than Participants: sides (left or right)
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
Number analyzed (sides (left or right)) | 20
sides (left or right) | 12

3. Primary Outcome: Facet Joint High Grade MRI Signal Change Concordance to Pain
Description: as for outcome 2
Time Frame: 2 years
Population: Two sides for each patient, for a total of 20 sides
Measure: Number; unit: sides (left or right)
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
sides (left or right) | 12

4. Primary Outcome: Facet Joint Any Grade of MRI Signal Change Concordance to Pain
Description: as for outcome 2
Time Frame: 2 years
Population: two sides for each patient, for a total of 20 sides
Measure: Number; unit: sides (Left or Right)
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
sides (Left or Right) | 12

5. Primary Outcome: Facet Joint High Grade FDG Activity Potential Effect on Management
Description: Number/percentage of subjects for whom high grade FDG scores would change clinical management
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
Participants | 8

6. Primary Outcome: Facet Joint All Grades of FDG Activity Potential Effect on Management
Description: Number/percentage of subjects for whom any grade FDG scores would change clinical management
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
Participants | 8

7. Primary Outcome: Facet Joint High Grade MRI Signal Change Potential Effect on Management
Description: Number/percentage of subjects for whom high grade MRI facet joint signal change would change clinical management
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
Participants | 8

8. Primary Outcome: Facet Joint Any Grade MRI Signal Change Potential Effect on Management
Description: Number/percentage of subjects for whom any grade MRI facet joint signal change would change clinical management
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PET/MR Recipients
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: 1 year
Description: No serious adverse events have been reported. No one is suspected to have a serious adverse event.
Arm/Group | PET/MR Recipients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET/MR Recipients (N=10)
IV site swelling (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT02921490/Prot_SAP_000.pdf